CLINICAL TRIAL: NCT00116779
Title: An Open-label, Randomized, Multi-center, Parallel Group Comparison of the Efficacy and Safety of Degarelix at Two Different Dosing Regimens in Patients With Prostate Cancer Dosed for Thirteen 28-day Cycles
Brief Title: A Parallel Group Comparison of the Efficacy and Safety of Degarelix at Two Different Dosing Regimens in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS14
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2009-03-20 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix 60mg (Experimental): Initial dose of 200 milligrams (40 milligrams per milliliter) of Degarelix on Day 0 (cycle 1) given by subcutaneous injection. Maintenance dose of 60 milligrams (20 milligrams per milliliter) of Degarelix given by subcutaneous injection every 28 days for cycles 2-13.
  Interventions: Drug: Degarelix
- Degarelix 80mg (Experimental): Initial dose of 200 milligrams (40 milligrams per milliliter) of Degarelix on Day 0 (cycle 1) given by subcutaneous injection. Maintenance dose of 80 milligrams (20 milligrams per milliliter) of Degarelix given by subcutaneous injection every 28 days for cycles 2 - 13.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Drug supplied as a powder to be dissolved in the solvent for solution for injection. Maintenance dose given in twelve 28-day cycles.
  Other Names: FE200486

SUMMARY:
The purpose of the study was to contribute, along with other such dose-finding studies, to the identification of the most effective treatment regimen for a one month depot injection of degarelix in the treatment of prostate cancer by a rapid and sustained suppression of testosterone.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following inclusion criteria before entry into the study.

* Has given written consent prior to any study-related activity is performed (a study-related activity is defined as any procedure that would not have been performed during the normal management of the patient).
* Histologically confirmed adenocarcinoma of the prostate (all stages), in whom endocrine treatment (except for neoadjuvant hormonal therapy) is indicated. This includes patients with rising PSA after having received radical prostatectomy (removal of the entire prostate and seminal vesicles) or radiotherapy with curative intention.
* Male patient aged 18 years or over.
* Has a baseline testosterone above the lower limit of normal range.
* Has an ECOG (Eastern Co-operative Oncology Group) score equal to or less than 2.
* Has a PSA value of greater than or equal to 2ng/mL.

Exclusion Criteria:

Any patient meeting one or more of the following exclusion criteria will not be entered into the study.

* Previous or present hormonal management of prostate cancer (surgical castration or other hormonal manipulation, e.g. GnRH agonists, GnRH antagonists, antiandrogens, estrogens). However, patients having undergone neoadjuvant hormonal therapy in conjunction with prostatectomy or radiotherapy with curative intention may be included so long as the hormonal therapy did not exceed a total duration of 6 months and was terminated at least 6 months prior to the Screening Visit.
* Currently or recently (within the last 12 weeks preceding the Screening Visit) under treatment with any other drug modifying testosterone level or function.
* Is considered to be a candidate for curative therapy, i.e., radical prostatectomy or radiotherapy within 6 months from Screening Visit.
* Has a history of severe asthma (defined as a need for daily treatment with oral or inhalation steroids to control the asthma), anaphylactic reactions, angioedema, angioneurotic edema or Quincke's Edema.
* Has hypersensitivity towards any component of the investigational products (degarelix or mannitol).
* Has history of other cancer within the last 5 years except for prostate cancer and surgically removed basal or squamous cell carcinoma of the skin.
* Has elevated serum ALT level more than three times above upper level of normal range or serum total bilirubin level above one and a half times above upper level of normal range as measured by the laboratory at the Screening Visit.
* Has known or suspect hepatic disease of any sort. Patients with liver disease are not to be enrolled in this study.
* Has other clinically significant laboratory abnormalities, which in the judgment of the investigator would interfere with the participation of the patient in this study or evaluation of study results.
* Has a clinically significant disorder (other than prostate cancer) or any other condition, including excessive alcohol or drug abuse, which may interfere with trial participation or which may affect the conclusion of the study as judged by the investigator.
* Has a mental incapacity or language barriers precluding adequate understanding or cooperation.
* Has received an investigational drug within the last 12 weeks preceding Screening Visit.
* Has previously participated in any degarelix study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (35):
- United States (26):
  - Urology Centers of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Advanced Urology Medical Center, Anaheim, California
  - South Orange County Medical Research Cnter, Laguna Woods, California
  - Pacific Clinical Research, Santa Monica, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Torrance, California
  - Urology Associate PC, Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - SW Florida Urological Associates, Fort Myers, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - RMD Clinical Reseach Institution LLC, Melrose Park, Illinois
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Regional Urology, Shreveport, Louisiana
  - Nevada Urology Associates, Reno, Nevada
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Hudson Valley Urology PC, Poughkeepsie, New York
  - The Urology Center, Greensboro, North Carolina
  - State College Urologic Association, State College, Pennsylvania
  - Univeristy Urological Research Institute, Providence, Rhode Island
  - Urology San Antonio Research, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Vermont, Dept of Surgery, South Burlington, Vermont
  - Virginia Urology Center, Richmond, Virginia
  - Office of Jeffrey Frankel, Seattle, Washington
  - Wyoming Research Foundation, Cheyenne, Wyoming
- Canada (9):
  - Southern Interior Medical Research Corporation, Kelowna, British Columbia
  - Dr. Cal Abdreau Research, Surrey, British Columbia
  - Can-Med Clinical Research, Inc., Victoria, British Columbia
  - Dr. Gary Steinhoff Clinical Research, Victoria, British Columbia
  - Valley Professional Center, Kentville, Nova Scotia
  - The Male and Female Health and Research Centers, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Burlington Professional Care, Burlington, Ontario
  - The Female/Male Health Centres, Oakville, Ontario

REFERENCES:
- [Result] Gittelman M, Pommerville PJ, Persson BE, Jensen JK, Olesen TK; Degarelix Study Group. A 1-year, open label, randomized phase II dose finding study of degarelix for the treatment of prostate cancer in North America. J Urol. 2008 Nov;180(5):1986-92. doi: 10.1016/j.juro.2008.07.033. Epub 2008 Sep 17. PMID 18801505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred and seventy-six patients were screened to identify the one hundred and twenty-seven patients who were eligible for randomization.
Groups:
- Degarelix 60mg: Initial dose of 200 milligrams of Degarelix on Day 0 (cycle 1) given by subcutaneous injection. Maintenance dose of 60 milligrams of Degarelix given by subcutaneous injection every 28 days for cycles 2-13.
- Degarelix 80mg: Initial dose of 200 milligrams of Degarelix on Day 0 (cycle 1) given by subcutaneous injection. Maintenance dose of 80 milligrams of Degarelix given by subcutaneous injection every 28 days for cycles 2 - 13.
Period: Overall Study
Arm/Group | Degarelix 60mg | Degarelix 80mg
Started | 63 (Randomized and treated; Intent-to-treat population) | 64 (Randomized and treated; intent-to-treat population)
Completed | 42 | 45
Not Completed | 21 | 19
Not completed — Adverse Event | 4 | 2
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Inadequate testosterone suppression | 7 | 9
Not completed — Physician Decision | 3 | 1
Not completed — Elevated PSA levels | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 60mg | Degarelix 80mg | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 54 | 55 | 109
Age Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.73) | 74.9 (9.55) | 74.9 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 63 | 64 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 4 | 18
  White | 48 | 59 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Curative Intent [Number; unit: participants] — A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    No | 41 | 40 | 81
    Yes | 22 | 24 | 46
Participant Counts by Gleason Score [Number; unit: participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    2-4 | 3 | 3 | 6
    5-6 | 19 | 22 | 41
    7-10 | 41 | 39 | 80
The Number of Participants at Each Stage of Prostate Cancer [Number; unit: participants] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 31 | 23 | 54
    Locally advanced | 5 | 9 | 14
    Metastatic | 15 | 9 | 24
    Not classifiable | 12 | 23 | 35
Body Mass Index [Mean (Full Range); unit: kilogram per square meter] — Body mass index is a measure of body fat based on height and weight.
  kilogram per square meter | 27.3 (4.1) [19.1 to 39.2] | 26.7 (3.98) [16.9 to 36.4] | 27 (4.03) [16.9 to 39.2]
Days Since Diagnosis of Prostate Cancer [Mean (Standard Deviation); unit: days] — The number of days passed since a diagnosis of prostate cancer was made for each participant.
  days | 1213 (1597) | 1256 (1550) | 1234 (1568)
Serum Prostate-Specific Antigen [Median (Full Range); unit: nanograms/milliliter] — Prostate-specific antigen (PSA) is a protein produced by the cells of the prostate gland. The PSA test measures the level of PSA in the blood. High PSA levels have a postive corrolation to prostate cancer.
  nanograms/milliliter | 12.7 [2.7 to 759] | 13.7 [1.6 to 1942] | 13.4 [1.6 to 1942]
Serum Testosterone level [Median (Full Range); unit: nanograms/milliliter] — Testosterone is a steroid hormone from the androgen group, and the principal male sex hormone. This test measures the amount of testosterone in the blood. Androgen deprivation is used to manage prostate cancer.
  nanograms/milliliter | 4.1 [1.51 to 11] | 4.23 [0.2 to 8.68] | 4.13 [0.2 to 11]
Weight [Mean (Standard Deviation); unit: Kilograms] — Mean of Participants Weight in Kilograms
  Kilograms | 83 (14.6) | 81.2 (12.7) | 82.1 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Testosterone <=0.5 Nanogram/Milliliter From Day 28 to Day 364
Description: Number of participants with all testosterone values <=0.5 nanogram/milliliter from Day 28 to Day 364
Time Frame: Day 28 to Day 364
Population: ITT population of patients who completed the study and had testosterone <=0.5 nanogram per milliliter at Day 28.
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 49 | 53
participants | 42 [73 to 94] | 41 [64 to 88]
Statistical Analysis 1: Comparison: Degarelix 60mg; Test type: Superiority or Other; Percentage of participants = 86, 95% CI [73 to 94] — The 95% confidence interval was calculated by Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 80mg; Test type: Superiority or Other; Percentage of participants = 77, 95% CI [64 to 88] — The 95% confidence interval was calculated by Clopper-Pearson method

2. Secondary Outcome: Number of Participants With Testosterone <= 0.5 Nanogram/Milliliter at Day 3.
Description: Testosterone levels checked at Day 3 to determine if the reduction in testosterone level occurs rapidly after dosing.
Time Frame: Day 3
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
participants | 54 [79 to 96] | 56 [78 to 95]
Statistical Analysis 1: Comparison: Degarelix 60mg; Test type: Superiority or Other; Percentage of participants = 90, 95% CI [79 to 96] — The 95% confidence interval was calculated by Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 80mg; Test type: Superiority or Other; Percentage of participants = 89, 95% CI [78 to 95] — The 95% confidence interval was calculated by Clopper-Pearson method
Statistical Analysis 3: Comparison: Degarelix 60mg vs Degarelix 80mg; Test type: Superiority or Other; p = 0.8413, Chi-squared

3. Primary Outcome: Number of Participants With Testosterone Level <= 0.5 Nanogram/Milliliter From Day 28 to Day 364 for Participants With Testosterone <= 0.5 Nanogram/Milliliter at Day 28
Description: Number of participants who maintained a testosterone level of <=0.5 nanogram/milliliter from Day 28 to Day 364.
Time Frame: Day 28 - Day 364
Population: ITT population of participants who completed the study and had a testosterone level of <=0.5 nanogram per milliliter at Day 28.
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 45 | 42
participants | 42 [82 to 99] | 41 [87 to 100]
Statistical Analysis 1: Comparison: Degarelix 60mg; Test type: Superiority or Other; Percentage of participants = 93, 95% CI [82 to 99] — The 95% confidence interval was calculated by Clopper-Pearson method
Statistical Analysis 2: Comparison: Degarelix 80mg; Test type: Superiority or Other; Percentage of participants = 98, 95% CI [87 to 100] — The 95% confidence interval was calculated by Clopper-Pearson method

4. Secondary Outcome: Days to 50 Percent and 90 Percent Reduction in Prostate-Specific Antigen
Description: Median number of days after the first dose of Degarelix when the Prostate-Specific Antigen levels fell to 50 percent and 90 percent of the baseline value.
Time Frame: Day 0 (post dose) to Day 364
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
days
  50 percent reduction (n=59, 59) | 14 [3 to 84] | 14 [1 to 56]
  90 percent reduction (n=45, 48) | 56 [28 to 168] | 56 [14 to 252]
Statistical Analysis 1: Comparison: Degarelix 60mg vs Degarelix 80mg; Time to 50% reduction; Test type: Superiority or Other; p = .904, Log Rank
Statistical Analysis 2: Comparison: Degarelix 60mg vs Degarelix 80mg; Days to 90% reduction; Test type: Superiority or Other; p = .778, Log Rank

5. Secondary Outcome: Days to Prostate-Specific Antigen Progression
Description: Median days to prostate-specific antigen increase of >= 50 percent and >= 5 nanograms/milliliter compared to nadir on two consecutive visits at least 2 weeks apart.
Time Frame: Day 0 (post dose) to Day 364
Population: ITT population. 5 patients in the 60 mg group and 4 patients in the 80 mg group had PSA progression.
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
days | 196 [107 to 280] | 154 [28 to 308]

6. Secondary Outcome: Median Di-Hydrotestosterone Levels At Various Study Timepoints
Description: Di-hydrotestosterone levels at baseline and days 1, 3, 7, 14
Time Frame: Baseline, Days 1, 3, 7, 14
Population: ITT population
Measure: Median (Full Range); unit: picogram / milliliter
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
picogram / milliliter
  Baseline (n=63, 64) | 360 [10 to 800] | 350 [48 to 810]
  Day 1 (n=62, 62) | 110 [37 to 350] | 120 [34 to 280]
  Day 3 (n=58, 63) | 56.5 [10 to 230] | 57 [10 to 150]
  Day 7 (n=58, 63) | 45.5 [20 to 150] | 52 [10 to 280]
  Day 14 (n=61, 61) | 37 [10 to 230] | 40 [10 to 430]

7. Secondary Outcome: Median Prostate-Specific Antigen Values at Various Study Timepoints
Description: Prostate-specific antigen levels at baseline and days 3, 14, 28, 84, and 364.
Time Frame: Baseline, Days 3, 14, 28, 84, 364
Population: ITT population
Measure: Median (Full Range); unit: nanogram / milliliter
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
nanogram / milliliter
  Baseline (n=63, 64) | 12.7 [2.7 to 759] | 13.7 [1.6 to 1942]
  Day 3 (n=60, 64) | 11.4 [2.1 to 1557] | 12.2 [1.3 to 1206]
  Day 14 (n=61, 63) | 6.4 [0.9 to 362] | 6.8 [0.9 to 182]
  Day 28 (n=61, 63) | 2.9 [0.3 to 28.8] | 3.6 [0.3 to 127]
  Day 84 (n=57, 54) | 0.8 [0 to 32.1] | 0.7 [0 to 104]
  Day 364 (n=42, 43) | 0.4 [0 to 12.8] | 0.2 [0 to 39.8]

8. Secondary Outcome: Median Luteinizing Hormone Levels at Various Study Timeframes
Description: Luteinizing hormone levels at baseline, and days 1, 3, 7, and 14.
Time Frame: Baseline, Days 1, 3, 7, 14
Population: ITT population
Measure: Median (Full Range); unit: international units / liter
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
international units / liter
  Baseline (n=63, 64) | 5.28 [1.22 to 25] | 5.33 [0.72 to 31]
  Day 1 (n=58, 61) | 0.915 [0.22 to 5.21] | 0.87 [0.035 to 5.64]
  Day 3 (n=59, 60) | 0.43 [0.035 to 2.05] | 0.425 [0.035 to 1.78]
  Day 7 (n=60, 61) | 0.41 [0.035 to 2.64] | 0.6 [0.035 to 7.35]
  Day 14 (n=61, 62) | 0.2 [0.035 to 3.5] | 0.37 [0.035 to 9.5]

9. Secondary Outcome: Median Testosterone Levels at Various Days During the Study
Description: Testosterone levels at baseline and days 1, 3, 7, 14 and 364
Time Frame: Baseline, Days 1,3,7,14,364
Population: ITT population
Measure: Median (Full Range); unit: nanograms / milliliter
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
nanograms / milliliter
  Baseline (n=63, 64) | 4.1 [1.51 to 11] | 4.23 [0.2 to 8.68]
  Day 1 (n=61, 63) | 0.56 [0.2 to 2.49] | 0.71 [0.12 to 2.98]
  Day 3 (n=60, 63) | 0.26 [0.13 to 0.67] | 0.31 [0.11 to 1.31]
  Day 7 (n=60, 64) | 0.18 [0.08 to 1.46] | 0.24 [0.07 to 3.98]
  Day 14 (n=61, 63) | 0.11 [0.04 to 2.19] | 0.14 [0.015 to 6.99]
  Day 364 (n=42, 43) | 0.07 [0.015 to 0.45] | 0.07 [0.015 to 0.32]

10. Secondary Outcome: Number of Participants With Abnormal Alanine Aminotransferase Values
Description: Participants whose alanine aminotransferase values were at levels above the normal range.
Time Frame: Day 1 through day 364
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 62 | 64
participants
  > upper limit and 3 times upper limit | 10 | 21
  Total abnormal (> upper limit) | 10 | 21
  Total normal (<=upper limit) | 52 | 43

11. Secondary Outcome: Number of Participants With Abnormal Aspartate Aminotransferase Values
Description: Participants with aspartate aminotransferase values that were above the normal range.
Time Frame: Day 1 - 364
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 62 | 64
participants
  > 3 times upper limit - 5 times upper limit | 0 | 1
  > upper limit - 3 times upper limit | 6 | 5
  Total Abnormal (> upper limit) | 6 | 6
  Total Normal (<= upper limit) | 56 | 58

12. Secondary Outcome: Number of Participants With Abnormal Total Bilirubin Values
Description: Participants with abnormal total bilirubin values
Time Frame: Day 1 - 364
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 62 | 64
participants
  >2 times upper limit | 0 | 1
  >1.5 times upper limit | 2 | 4
  > upper limit - 1.5 times upper limit | 12 | 9
  Total abnormal (> upper limit) | 14 | 14
  Total normal (<=upper limit) | 48 | 50

13. Secondary Outcome: Participants With Markedly Abnormal Changes in Vital Signs or Body Weight
Description: Vital sign and body weight values at the end of the trial are compared to baseline values. The table represents the number of participants in each group with normal baseline values and markedly abnormal end-of-study values.
Time Frame: Day 364
Population: ITT population. Diastolic blood pressure n=63,63 Pulse n=63,60 Systolic blood pressure n=63,64 Weight n=55,61
Measure: Number; unit: participants
Arm/Group | Degarelix 60mg | Degarelix 80mg
Number analyzed (Participants) | 63 | 64
participants
  Diastolic blood pressure <= 50 and decrease >= 15 | 7 | 5
  Diastolic blood pressure >= 105 and increase >= 15 | 1 | 2
  Pulse <=50 and decrease of >=15 | 2 | 5
  Pulse >=120 and increase of >=15 | 0 | 0
  Systolic blood pressure <=90 and decrease >=20 | 5 | 5
  Systolic blood pressure >=180 and increase >=20 | 6 | 7
  Weight decrease of >=7 percent | 2 | 3
  Weight increase of >= 7 percent | 7 | 4

ADVERSE EVENTS:
Arm/Group | Degarelix 60mg | Degarelix 80mg
Serious Adverse Events (participants affected / at risk) | 9 | 6
Other Adverse Events (participants affected / at risk) | 55 | 52
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 60mg | Degarelix 80mg
Myocardial infarction (Cardiac disorders) | 1/63 (1) | 1/64 (1)
Acute coronary syndrome (Cardiac disorders) | 1/63 (1) | 0/64 (0)
Acute myocardial infarction (Cardiac disorders) | 0/63 (0) | 1/64 (1)
Coronary artery disease (Cardiac disorders) | 0/63 (0) | 1/64 (1)
Constipation (Gastrointestinal disorders) | 1/63 (1) | 0/64 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0/63 (0) | 1/64 (1)
Injection site urticaria (General disorders) | 1/63 (1) | 0/64 (0)
Cholelithiasis (Hepatobiliary disorders) | 0/63 (0) | 1/64 (1)
Pneumonia (Infections and infestations) | 1/63 (1) | 1/64 (1)
Orchitis (Infections and infestations) | 1/63 (1) | 0/64 (0)
Perirectal abscess (Infections and infestations) | 1/63 (1) | 0/64 (0)
Pseudomembranous colitis (Infections and infestations) | 1/63 (1) | 0/64 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1/63 (1) | 0/64 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/63 (1) | 0/64 (0)
Grand mal convulsion (Nervous system disorders) | 1/63 (1) | 0/64 (0)
Transient ischaemic attack (Nervous system disorders) | 1/63 (1) | 0/64 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0/63 (0) | 1/64 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/63 (1) | 0/64 (0)
Deep vein thrombosis (Vascular disorders) | 1/63 (1) | 0/64 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 60mg | Degarelix 80mg
Anaemia (Blood and lymphatic system disorders) | 3/63 (3) | 2/64 (2)
Constipation (Gastrointestinal disorders) | 4/63 (4) | 4/64 (4)
Diarrhoea (Gastrointestinal disorders) | 3/63 (3) | 2/64 (2)
Nausea (Gastrointestinal disorders) | 3/63 (4) | 2/64 (2)
Fatigue (General disorders) | 10/63 (12) | 15/64 (18)
Injection site pain (General disorders) | 4/63 (5) | 5/64 (9)
Asthenia (General disorders) | 2/63 (2) | 4/64 (5)
Nasopharyngitis (Infections and infestations) | 7/63 (10) | 7/64 (7)
Upper respiratory tract infection (Infections and infestations) | 1/63 (1) | 5/64 (6)
Urinary tract infection (Infections and infestations) | 3/63 (4) | 2/64 (3)
Lower respiratory tract infection (Infections and infestations) | 1/63 (1) | 3/64 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 3/63 (3) | 0/64 (0)
Weight increased (Investigations) | 4/63 (4) | 4/64 (4)
Gamma-glutamyltransferase increased (Investigations) | 1/63 (2) | 3/64 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/63 (4) | 4/64 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2/63 (2) | 5/64 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/63 (0) | 3/64 (4)
Dizziness (Nervous system disorders) | 7/63 (11) | 6/64 (7)
Insomnia (Psychiatric disorders) | 2/63 (2) | 5/64 (6)
Anxiety (Psychiatric disorders) | 3/63 (3) | 1/64 (2)
Nocturia (Renal and urinary disorders) | 1/63 (1) | 7/64 (7)
Dysuria (Renal and urinary disorders) | 3/63 (3) | 3/64 (4)
Micturition urgency (Renal and urinary disorders) | 1/63 (1) | 4/64 (5)
Pollakiuria (Renal and urinary disorders) | 4/63 (4) | 1/64 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 4/63 (4) | 6/64 (6)
Gynaecomastia (Reproductive system and breast disorders) | 3/63 (3) | 3/64 (4)
Rash (Skin and subcutaneous tissue disorders) | 3/63 (4) | 3/64 (3)
Hot flush (Vascular disorders) | 24/63 (26) | 31/64 (37)
Hypertension (Vascular disorders) | 4/63 (4) | 4/64 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of ublication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.